CLINICAL TRIAL: NCT00682552
Title: Evaluation of Initial High Risk Human Papillomavirus (HR-HPV) Viral Load as Predictive Marker for Cervical Intraepithelial Neoplasia Grade 1 (CIN1) Persistence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-A01336-48; 2007-31
Record Dates: First submitted 2008-05-19; First posted 2008-05-22 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): A cervico-vaginal cervical smear will be realized before every colposcopique examination.
  A new cervical taking for the search(research) and the detection of the HPV 16 and 18 will be realized.
  Interventions: Procedure: A cervico-vaginal cervical smear

INTERVENTIONS:
Procedure: A cervico-vaginal cervical smear — 12 and 18 months after inclusion, a cervico-vaginal cervical smear will be realized and a new examination colposcopique with a new cervical taking for the search(research) and the detection of the HPV 16 and 18.

SUMMARY:
Relationship between HPV infection and cervical cancer is well established. Among the HPV types identified to date, 15 are classified as high risk HPV (HR-HPV). Detection of HR-HPV has been proposed to optimize cervical cancer screening.

DETAILED DESCRIPTION:
A prospective detection and quantification of HR-HPV in patients with proven CIN1 will be performed. Relationship between HR-HPV initial viral load and the CIN1 persistence will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The women whose last one FCV of screening put in evidence a LIEBG of the neck of the womb having been confirmed by the colposcopie.
* The inclusive patients will be of more than 18 years old. All the patients will be profitable of a regime of Social Security.

Exclusion Criteria:

* The patients whose result of the colposcopie is clashing with that of the FCV of initial screening (normal collar, LIEHG or the other one).
* The patients having an antecedent of DREGS of the neck of the womb, that this one was or not handled
* The patients having had a hysterectomy.
* The patients incapable to receive the information enlightened on the progress and the objectives of the study
* The patients not having signed enlightened assent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The detection and the quantification of the DNA of the human oncogènes papillomavirus of type 16 and 18 | 48 months

SECONDARY OUTCOMES:
The detection of the markers of the integration of the genome of the human oncogenes papillomavirus (targeted at the gene E2) | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier CARCOPINO, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Hopital Nord- Service de gynécologie-obstétrique, Marseille, France